CLINICAL TRIAL: NCT06050278
Title: Prospective Evaluation of Single Cell Mutations in a Panel of Known Oncogenes in NSCLC Surgical Specimens (TAP-NSCLC)
Brief Title: Prospective Evaluation of Single Cell Mutations in a Panel of Known Oncogenes in NSCLC Surgical Specimens
Acronym: TAP-NSCLC
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: TAP-NSCLC
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples obtained from surgical treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tapestry technology — The study involves the immediate freezing and preservation in liquid nitrogen of a tumor histological sample from surgical resection, obtained from the operating room, within one hour of removal. Surgery is part of the normal clinical practice of patients with lung cancer.

SUMMARY:
The goal of this observational study is to evaluate the feasibility of a single cell mutation research method in a panel of known oncogenes, using the Tapestri method. Tissue samples will be obtained after surgical treatment in patients with I-II-III stage NSCLC.

DETAILED DESCRIPTION:
NSCLC is a particularly heterogeneous disease with different genetic alterations in oncogenes 'drivers', responsible for the development and progression of the disease. In most cases all these anomalies represent clonal mutations in all neoplastic cells. However, several sub-clonal genetic alterations were identified in some multi-regional sequencing studies, demonstrating an intra-tumor heterogeneity. Tracing the clonal architecture of the disease and also the temporal order of the various mutations appearance, would bring two benefits:

1. prioritize the molecular targets
2. identify evolutionary trajectories associated with the outcome of therapies and survival, useful to stratify patients considering the likelihood and the duration of response For the bioinformatic data analyses will be used the Tapestri MissionBio pipeline.

Given the limited number of patients that can be included in the study (10 patients), no statistical analyzes will be performed. Results will be presented thorugh narrative reports for each patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years old.
* histological diagnosis of NSCLC technically operable following multidisciplinary discussion
* informed consent freely granted and obtained before the start of the study

Exclusion Criteria:

* age under 18 years old
* unconfirmed NSCLC histological diagnosis
* medical treatment with neoadjuvant purposes
* absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects older than 18 years old, male and female, with histological diagnosis of NSCLC technically operable following multisciplinary discussion.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Tapestri success rate | 6 months
  Evaluation of the feasibility of a single cell mutation search method in a panel of known oncogenes, using Tapestri technology, in tumor tissue obtained from stage I-II-III NSCLC patients after surgical treatment planned in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: CSR
Time Frame: After publication
Access Criteria: Upon request